CLINICAL TRIAL: NCT05046912
Title: Exploring the Impact of Online Yoga on Outcome and Recovery in People With Psychosis.
Brief Title: Online Yoga and the Impact on Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021021
Record Dates: First submitted 2021-06-15; First posted 2021-09-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2021-09

CONDITIONS: Psychosis
Keywords: Psychosis; Yoga; Mindfulness; Recovery; Online
MeSH Terms: conditions — Psychotic Disorders | interventions — Yoga; Mindfulness

STUDY DESIGN:
Intervention Model Description: Clinical and non-clinical participants will be assigned to either a yoga or mindfulness condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical (Experimental): Clinical participants with a primary diagnosis of psychosis or related disorder.
  Interventions: Behavioral: Yoga; Behavioral: Mindfulness
- Non-clinical (Active Comparator): Non-clinical participants with no mental health diagnoses.
  Interventions: Behavioral: Yoga; Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Yoga — 8 weeks of online weekly yoga or chair yoga class
Behavioral: Mindfulness — 8 weeks of online weekly mindfulness class

SUMMARY:
Yoga and mindfulness are considered complementary and alternative healthcare options that involve breathing techniques, relaxation, and bodily postures (yoga only). Research has shown a positive effect of these on depression, quality of life, and other symptoms of psychosis. As an 8-week pilot study, the goal is to offer yoga and/or mindfulness online and to explore the effect on recovery and quality of life for people with psychosis.

DETAILED DESCRIPTION:
Psychosis impacts about 3% of Canadians at any given time. People with psychosis can experience a combination of positive (e.g., delusions; hallucinations), negative (e.g., amotivation; reduced social activity), or cognitive symptoms (e.g., poorer memory; executive functioning). Positive symptoms are managed via antipsychotic medication and therapeutic support; cognitive symptoms can be targeted via cognitive remediation therapy. For negative symptoms, especially those idiopathic, there are still no effective care options. Yoga is a complementary and alternative medicine (CAM) encompassing health modalities of Eastern cultures, it involves breathing techniques, relaxation, and bodily postures. Research has shown that yoga can improve levels of depression and quality of life, and even attenuate negative symptoms. Given the extensive health care expenditures and unmet care needs for negative symptoms, there is a growing need to consider CAMs, such as yoga, and accessibility of CAMs via online methods. As a pioneering study, this proposed pilot study aims to explore the effect of an 8-week (i.e., 8 sessions) online yoga program on recovery/outcome, with a focus on negative symptoms, for people with psychosis. The investigators aim to recruit 24 people with psychosis and randomly assign them to either the yoga (n=12) or a mindfulness group (n=12); mindfulness, in essence, is yoga without the physical aspect (i.e., poses). The investigators hypothesize that yoga will improve quality of life and attenuate symptom severity, with a larger effect on negative symptoms, above the effect of mindfulness. A nonclinical sample (n=12) will also be recruited to examine feasibility and for feedback purposes.

ELIGIBILITY:
Inclusion Criteria:

For clinical participants:

* primary diagnosis of a schizophrenia-spectrum disorder (schizophrenia, schizophreniform, schizoaffective) or related psychotic disorder (delusional, brief psychotic, paraphrenia, bipolar with psychotic features, major-depressive with psychotic features)
* access to protected internet (i.e., home internet plugged or password protected wireless)
* adequate space to do yoga (e.g., at least 2 feet around each side of the yoga mat)
* able to speak and read English
* competent and able to offer voluntary informed consent to participate

For non-clinical participants (healthy controls):

* not diagnosed with or received care for any mental illness
* access to protected internet (i.e., home internet plugged or password protected wireless)
* adequate space to do yoga (e.g., at least 2 feet around each side of the yoga mat)
* able to speak and read English
* competent and able to offer voluntary informed consent to participate

Exclusion Criteria:

For clinical participants:

* not clinically stable; that is, major change in primary medication (e.g., switching or stopping antipsychotic) or hospitalisation within the past 4 weeks prior to first contact
* currently with a physical ailment that restricts light movement exercises for yoga or chair yoga

For non-clinical participants (healthy controls):

* have a first-degree relative with psychosis (schizophrenia, schizo-affective, schizophreniform, paraphrenia, brief psychotic, delusional, or bipolar or major depressive disorder with psychotic features)
* had a substance or alcohol abuse/dependence in the past 6 months
* currently with a physical ailment that restricts light movement exercises for yoga or chair yoga

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-11-05 (Estimated); Study Completion 2022-11-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on the Clinical Outcomes in Routine Evaluation (CORE-10) scale at week 4 | Baseline and Week 4
  The CORE-10 is a self-reported instrument measuring levels of psychological distress in the past week. Possible scores range from 0 (not at all) to 4 (most or all of the time). Higher score = worse outcome. Change = (week 4 - baseline).
Change from baseline on the Clinical Outcomes in Routine Evaluation (CORE-10) scale at week 8 | Baseline and Week 8
  The CORE-10 is a self-reported instrument measuring levels of psychological distress in the past week. Possible scores range from 0 (not at all) to 4 (most or all of the time). Higher score = worse outcome. Change = (week 8 - baseline).
Change from baseline on the Clinical Outcomes in Routine Evaluation (CORE-10) scale at week 12 | Baseline and Week 12
  The CORE-10 is a self-reported instrument measuring levels of psychological distress in the past week. Possible scores range from 0 (not at all) to 4 (most or all of the time). Higher score = worse outcome. Change = (week 12 - baseline).
Change from baseline on the Clinical Outcomes in Routine Evaluation (CORE-10) scale at 6 months | Baseline and 6 Months
  The CORE-10 is a self-reported instrument measuring levels of psychological distress in the past week. Possible scores range from 0 (not at all) to 4 (most or all of the time). Higher score = worse outcome. Change = (6 month - baseline).
Change from baseline on the Positive and Negative Syndrome Scale for Schizophrenia (PANSS) scale at 4 weeks | Baseline and Week 4
  The PANSS is a clinician-rated, semi-structured interview assessing schizophrenia symptom severity over the past week. Possible scores range from 1 (absent) to 7 (extreme). Higher score = worse outcome. Change = (week 4 - baseline).
Change from baseline on the Positive and Negative Syndrome Scale for Schizophrenia (PANSS) scale at 8 weeks | Baseline and Week 8
  The PANSS is a clinician-rated, semi-structured interview assessing schizophrenia symptom severity over the past week. Possible scores range from 1 (absent) to 7 (extreme). Higher score = worse outcome. Change = (week 8 - baseline).
Change from baseline on the Positive and Negative Syndrome Scale for Schizophrenia (PANSS) scale at 12 weeks | Baseline and Week 12
  The PANSS is a clinician-rated, semi-structured interview assessing schizophrenia symptom severity over the past week. Possible scores range from 1 (absent) to 7 (extreme). Higher score = worse outcome. Change = (week 12 - baseline).
Change from baseline on the Positive and Negative Syndrome Scale for Schizophrenia (PANSS) scale at 6 months | Baseline and 6 Months
  The PANSS is a clinician-rated, semi-structured interview assessing schizophrenia symptom severity over the past week. Possible scores range from 1 (absent) to 7 (extreme). Higher score = worse outcome. Change = (6 month - baseline).
Change from baseline on the Questionnaire about the Process of Recovery - Version 2 (QPR-2) scale at week 4 | Baseline and Week 4
  The QPR-2 is a self-reported instrument assessing levels of recovery over the past week. Scores range from 0 (disagree strongly) to 4 (agree strongly). Higher score = better outcome. Change = (week 4 - baseline).
Change from baseline on the Questionnaire about the Process of Recovery - Version 2 (QPR-2) scale at week 8 | Baseline and Week 8
  The QPR-2 is a self-reported instrument assessing levels of recovery over the past week. Scores range from 0 (disagree strongly) to 4 (agree strongly). Higher score = better outcome. Change = (week 8 - baseline).
Change from baseline on the Questionnaire about the Process of Recovery - Version 2 (QPR-2) scale at week 12 | Baseline and Week 12
  The QPR-2 is a self-reported instrument assessing levels of recovery over the past week. Scores range from 0 (disagree strongly) to 4 (agree strongly). Higher score = better outcome. Change = (week 12 - baseline).
Change from baseline on the Questionnaire about the Process of Recovery - Version 2 (QPR-2) scale at 6 months | Baseline and 6 Months
  The QPR-2 is a self-reported instrument assessing levels of recovery over the past week. Scores range from 0 (disagree strongly) to 4 (agree strongly). Higher score = better outcome. Change = (6 months - baseline).
Change from baseline on the Self-Evaluation of Negative Symptoms (SNS) scale at week 4 | Baseline and Week 4
  The SNS is a self-reported instrument assessing negative symptom severity over the past week. Possible answers are strongly agree, somewhat agree, strongly disagree. Higher score = worse outcome. Change = (week 4 - baseline).
Change from baseline on the Self-Evaluation of Negative Symptoms (SNS) scale at week 8 | Baseline and Week 8
  The SNS is a self-reported instrument assessing negative symptom severity over the past week. Possible answers are strongly agree, somewhat agree, strongly disagree. Higher score = worse outcome. Change = (week 8 - baseline).
Change from baseline on the Self-Evaluation of Negative Symptoms (SNS) scale at week 12 | Baseline and Week 12
  The SNS is a self-reported instrument assessing negative symptom severity over the past week. Possible answers are strongly agree, somewhat agree, strongly disagree. Higher score = worse outcome. Change = (week 12 - baseline).
Change from baseline on the Self-Evaluation of Negative Symptoms (SNS) scale at 6 months | Baseline and 6 Months
  The SNS is a self-reported instrument assessing negative symptom severity over the past week. Possible answers are strongly agree, somewhat agree, strongly disagree. Higher score = worse outcome. Change = (6 months - baseline).
Change from baseline on the Birchwood Insight Scale (BIS) scale at week 4 | Baseline and Week 4
  The BIS is a self-reported instrument assessing levels of insight without a specific time period. Possible answers are agree, disagree, unsure. Higher score = better outcome. Change = (week 4 - baseline).
Change from baseline on the Birchwood Insight Scale (BIS) scale at week 8 | Baseline and Week 8
  The BIS is a self-reported instrument assessing levels of insight without a specific time period. Possible answers are agree, disagree, unsure. Higher score = better outcome. Change = (week 8 - baseline).
Change from baseline on the Birchwood Insight Scale (BIS) scale at week 12 | Baseline and Week 12
  The BIS is a self-reported instrument assessing levels of insight without a specific time period. Possible answers are agree, disagree, unsure. Higher score = better outcome. Change = (week 12 - baseline).
Change from baseline on the Birchwood Insight Scale (BIS) scale at 6 months | Baseline and 6 Months
  The BIS is a self-reported instrument assessing levels of insight without a specific time period. Possible answers are agree, disagree, unsure. Higher score = better outcome. Change = (6 months - baseline).
Change from baseline on the Short Warwick Edinburgh Mental Well-Being Scale (SWEMWBS) scale at week 4 | Baseline and Week 4
  The SWEMWBS is a self-reported instrument assessing levels of overall mental well-being over the past 2 weeks. Possible scores range from 1 (none of the time) to 5 (all of the time). Higher score = better outcome. Change = (week 4 - baseline).
Change from baseline on the Short Warwick Edinburgh Mental Well-Being Scale (SWEMWBS) scale at week 8 | Baseline and Week 8
  The SWEMWBS is a self-reported instrument assessing levels of overall mental well-being over the past 2 weeks. Possible scores range from 1 (none of the time) to 5 (all of the time). Higher score = better outcome. Change = (week 8 - baseline).
Change from baseline on the Short Warwick Edinburgh Mental Well-Being Scale (SWEMWBS) scale at week 12 | Baseline and Week 12
  The SWEMWBS is a self-reported instrument assessing levels of overall mental well-being over the past 2 weeks. Possible scores range from 1 (none of the time) to 5 (all of the time). Higher score = better outcome. Change = (week 12 - baseline).
Change from baseline on the Short Warwick Edinburgh Mental Well-Being Scale (SWEMWBS) scale at 6 months | Baseline and 6 Months
  The SWEMWBS is a self-reported instrument assessing levels of overall mental well-being over the past 2 weeks. Possible scores range from 1 (none of the time) to 5 (all of the time). Higher score = better outcome. Change = (6 months - baseline).
Change from baseline on the Modified Global Assessment of Functioning - Revised (M-GAF(R)) scale at week 4 | Baseline and Week 4
  The M-GAF(R) is a clinician-rated instrument assessing overall level of functioning over the past month. Score ranges from 1 (severely impaired) to 100 (superior functioning). Higher score = better outcome. Change = (week 4 - baseline).
Change from baseline on the Modified Global Assessment of Functioning - Revised (M-GAF(R)) scale at week 8 | Baseline and Week 8
  The M-GAF(R) is a clinician-rated instrument assessing overall level of functioning over the past month. Score ranges from 1 (severely impaired) to 100 (superior functioning). Higher score = better outcome. Change = (week 8 - baseline).
Change from baseline on the Modified Global Assessment of Functioning - Revised (M-GAF(R)) scale at week 12 | Baseline and Week 12
  The M-GAF(R) is a clinician-rated instrument assessing overall level of functioning over the past month. Score ranges from 1 (severely impaired) to 100 (superior functioning). Higher score = better outcome. Change = (week 12 - baseline).
Change from baseline on the Modified Global Assessment of Functioning - Revised (M-GAF(R)) scale at 6 months | Baseline and 6 Months
  The M-GAF(R) is a clinician-rated instrument assessing overall level of functioning over the past month. Score ranges from 1 (severely impaired) to 100 (superior functioning). Higher score = better outcome. Change = (6 months - baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bodnar, PhD, Principal Investigator — The Royal Ottawa Mental Health Centre
Locations (1):
- The Royal Ottawa Mental Heatlh Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson G. Internet-Delivered Psychological Treatments. Annu Rev Clin Psychol. 2016;12:157-79. doi: 10.1146/annurev-clinpsy-021815-093006. Epub 2015 Dec 11. PMID 26652054
- [Background] Andersson G, Titov N, Dear BF, Rozental A, Carlbring P. Internet-delivered psychological treatments: from innovation to implementation. World Psychiatry. 2019 Feb;18(1):20-28. doi: 10.1002/wps.20610. PMID 30600624
- [Background] Aust J, Bradshaw T. Mindfulness interventions for psychosis: a systematic review of the literature. J Psychiatr Ment Health Nurs. 2017 Feb;24(1):69-83. doi: 10.1111/jpm.12357. Epub 2016 Dec 8. PMID 27928859
- [Background] Bartels SJ, Clark RE, Peacock WJ, Dums AR, Pratt SI. Medicare and medicaid costs for schizophrenia patients by age cohort compared with costs for depression, dementia, and medically ill patients. Am J Geriatr Psychiatry. 2003 Nov-Dec;11(6):648-57. doi: 10.1176/appi.ajgp.11.6.648. PMID 14609805
- [Background] Jayaram N, Varambally S, Behere RV, Venkatasubramanian G, Arasappa R, Christopher R, Gangadhar BN. Effect of yoga therapy on plasma oxytocin and facial emotion recognition deficits in patients of schizophrenia. Indian J Psychiatry. 2013 Jul;55(Suppl 3):S409-13. doi: 10.4103/0019-5545.116318. PMID 24049210
- [Background] Birchwood M, Smith J, Drury V, Healy J, Macmillan F, Slade M. A self-report Insight Scale for psychosis: reliability, validity and sensitivity to change. Acta Psychiatr Scand. 1994 Jan;89(1):62-7. doi: 10.1111/j.1600-0447.1994.tb01487.x. PMID 7908156
- [Background] Chang CK, Hayes RD, Perera G, Broadbent MT, Fernandes AC, Lee WE, Hotopf M, Stewart R. Life expectancy at birth for people with serious mental illness and other major disorders from a secondary mental health care case register in London. PLoS One. 2011;6(5):e19590. doi: 10.1371/journal.pone.0019590. Epub 2011 May 18. PMID 21611123
- [Background] Cramer H, Lauche R, Haller H, Langhorst J, Dobos G. Mindfulness- and Acceptance-based Interventions for Psychosis: A Systematic Review and Meta-analysis. Glob Adv Health Med. 2016 Jan;5(1):30-43. doi: 10.7453/gahmj.2015.083. Epub 2016 Jan 1. PMID 26937312
- [Background] Dollfus S, Mach C, Morello R. Self-Evaluation of Negative Symptoms: A Novel Tool to Assess Negative Symptoms. Schizophr Bull. 2016 May;42(3):571-8. doi: 10.1093/schbul/sbv161. Epub 2015 Nov 12. PMID 26564898
- [Background] Duraiswamy G, Thirthalli J, Nagendra HR, Gangadhar BN. Yoga therapy as an add-on treatment in the management of patients with schizophrenia--a randomized controlled trial. Acta Psychiatr Scand. 2007 Sep;116(3):226-32. doi: 10.1111/j.1600-0447.2007.01032.x. PMID 17655565
- [Background] Foussias G, Agid O, Fervaha G, Remington G. Negative symptoms of schizophrenia: clinical features, relevance to real world functioning and specificity versus other CNS disorders. Eur Neuropsychopharmacol. 2014 May;24(5):693-709. doi: 10.1016/j.euroneuro.2013.10.017. Epub 2013 Nov 11. PMID 24275699
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Kolbaek P, Blicher AB, Buus CW, Feller SG, Holm T, Dines D, O'Leary KM, Sorensen RS, Opler M, Correll CU, Mors O, Bech P, Ostergaard SD. Inter-rater reliability of ratings on the six-item Positive and Negative Syndrome Scale (PANSS-6) obtained using the Simplified Negative and Positive Symptoms Interview (SNAPSI). Nord J Psychiatry. 2018 Aug;72(6):431-436. doi: 10.1080/08039488.2018.1492014. Epub 2018 Jul 24. PMID 30037286
- [Background] Krause M, Zhu Y, Huhn M, Schneider-Thoma J, Bighelli I, Nikolakopoulou A, Leucht S. Antipsychotic drugs for patients with schizophrenia and predominant or prominent negative symptoms: a systematic review and meta-analysis. Eur Arch Psychiatry Clin Neurosci. 2018 Oct;268(7):625-639. doi: 10.1007/s00406-018-0869-3. Epub 2018 Jan 24. PMID 29368205
- [Background] Leucht S. Measurements of response, remission, and recovery in schizophrenia and examples for their clinical application. J Clin Psychiatry. 2014;75 Suppl 1:8-14. doi: 10.4088/JCP.13049su1c.02. PMID 24581453
- [Background] Leucht S, Leucht C, Huhn M, Chaimani A, Mavridis D, Helfer B, Samara M, Rabaioli M, Bacher S, Cipriani A, Geddes JR, Salanti G, Davis JM. Sixty Years of Placebo-Controlled Antipsychotic Drug Trials in Acute Schizophrenia: Systematic Review, Bayesian Meta-Analysis, and Meta-Regression of Efficacy Predictors. Am J Psychiatry. 2017 Oct 1;174(10):927-942. doi: 10.1176/appi.ajp.2017.16121358. Epub 2017 May 25. PMID 28541090
- [Background] Ostergaard SD, Lemming OM, Mors O, Correll CU, Bech P. PANSS-6: a brief rating scale for the measurement of severity in schizophrenia. Acta Psychiatr Scand. 2016 Jun;133(6):436-44. doi: 10.1111/acps.12526. Epub 2015 Nov 12. PMID 26558537
- [Background] Ostergaard SD, Opler MGA, Correll CU. Bridging the Measurement Gap Between Research and Clinical Care in Schizophrenia: Positive and Negative Syndrome Scale-6 (PANSS-6) and Other Assessments Based on the Simplified Negative and Positive Symptoms Interview (SNAPSI). Innov Clin Neurosci. 2017 Dec 1;14(11-12):68-72. PMID 29410939
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Spijkerman MP, Pots WT, Bohlmeijer ET. Effectiveness of online mindfulness-based interventions in improving mental health: A review and meta-analysis of randomised controlled trials. Clin Psychol Rev. 2016 Apr;45:102-14. doi: 10.1016/j.cpr.2016.03.009. Epub 2016 Apr 1. PMID 27111302
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Uebelacker L, Dufour SC, Dinerman JG, Walsh SL, Hearing C, Gillette LT, Deckersbach T, Nierenberg AA, Weinstock L, Sylvia LG. Examining the Feasibility and Acceptability of an Online Yoga Class for Mood Disorders: A MoodNetwork Study. J Psychiatr Pract. 2018 Jan;24(1):60-67. doi: 10.1097/PRA.0000000000000286. PMID 29320386
- [Background] van der Krieke L, Wunderink L, Emerencia AC, de Jonge P, Sytema S. E-mental health self-management for psychotic disorders: state of the art and future perspectives. Psychiatr Serv. 2014 Jan 1;65(1):33-49. doi: 10.1176/appi.ps.201300050. PMID 24129842
- [Background] Vancampfort D, Vansteelandt K, Scheewe T, Probst M, Knapen J, De Herdt A, De Hert M. Yoga in schizophrenia: a systematic review of randomised controlled trials. Acta Psychiatr Scand. 2012 Jul;126(1):12-20. doi: 10.1111/j.1600-0447.2012.01865.x. Epub 2012 Apr 6. PMID 22486714
- [Background] Varambally S, Gangadhar BN. Yoga: a spiritual practice with therapeutic value in psychiatry. Asian J Psychiatr. 2012 Jun;5(2):186-9. doi: 10.1016/j.ajp.2012.05.003. Epub 2012 May 18. PMID 22813667
- [Background] Varambally S, Gangadhar BN, Thirthalli J, Jagannathan A, Kumar S, Venkatasubramanian G, Muralidhar D, Subbakrishna DK, Nagendra HR. Therapeutic efficacy of add-on yogasana intervention in stabilized outpatient schizophrenia: Randomized controlled comparison with exercise and waitlist. Indian J Psychiatry. 2012 Jul;54(3):227-32. doi: 10.4103/0019-5545.102414. PMID 23226845
- [Background] Visceglia E, Lewis S. Yoga therapy as an adjunctive treatment for schizophrenia: a randomized, controlled pilot study. J Altern Complement Med. 2011 Jul;17(7):601-7. doi: 10.1089/acm.2010.0075. PMID 21711202
- [Background] Wolever RQ, Bobinet KJ, McCabe K, Mackenzie ER, Fekete E, Kusnick CA, Baime M. Effective and viable mind-body stress reduction in the workplace: a randomized controlled trial. J Occup Health Psychol. 2012 Apr;17(2):246-258. doi: 10.1037/a0027278. Epub 2012 Feb 20. PMID 22352291